CLINICAL TRIAL: NCT07349121
Title: Concomitant Left Atrial Appendage Closure and Pulsed Field Ablation - Europe, Middle East and Africa [OPTION-EMEA]
Brief Title: OPTION-EMEA Clinical Trial
Acronym: OPTION-EMEA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S2605
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF); Stroke Prevention in Patients With Atrial Fibrillation; Left Atrial Appendage Closure; Pulsed Field Ablation; Atrial Fibrillation Ablation Procedure; Concomitant Procedures
Keywords: WATCHMAN; FARAPULSE; Concomitant; PFA; LAAC
MeSH Terms: conditions — Atrial Fibrillation | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm study (Other): Subjects who meet eligibility criteria will undergo AF ablation and left atrial appendage closure using the FARAPULSE PFA system and WATCHMAN FLX Pro or WATCHMAN FLX during one interventional case.
  Interventions: Device: Concomitant pulsed field ablation (PFA) and left atrial appendage closure (LAAC) during one interventional case; Procedure: Concomitant Pulsed Field Ablation and Left Atrial Appendage Closure

INTERVENTIONS:
Device: Concomitant pulsed field ablation (PFA) and left atrial appendage closure (LAAC) during one interventional case — left atrial appendage closure
Procedure: Concomitant Pulsed Field Ablation and Left Atrial Appendage Closure — FARAPULSE PFA and WATCHMAN FLX Pro or WATCHMAN FLX in one interventional case.

SUMMARY:
The OPTION-EMEA post-market study is intended to gather real world clinical data for patients undergoing AF ablation with the FARAPULSE™ Pulsed Field Ablation (PFA) System and subsequent left atrial appendage closure (LAAC) with a WATCHMAN FLX™ Pro or WATCHMAN FLX device during one interventional case.

The study will include patients that are clinically indicated for atrial fibrillation (AF) ablation using the FARAPULSE PFA System and for left atrial appendage closure (LAAC) treatment using a WATCHMAN FLX Pro or WATCHMAN FLX device as part of the patient's standard of care determined by their doctor's medical judgement.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically indicated for treatment with both the FARAPULSE™ PFA system and with WATCHMAN FLX™ Pro or WATCHMAN FLX™ for LAAC, per physician medical judgement and as per hospitals' standard of care.
2. Subjects who are willing and able to provide informed consent.
3. Subjects who are willing and able to participate in all testing associated with this clinical study at an approved investigational center.
4. Subjects whose age is 18 years or above, or who are of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

1. Subjects who underwent prior AF ablation procedure.
2. Subjects with atrial fibrillation that is secondary to electrolyte imbalance, thyroid disease, alcohol, or other reversible / non-cardiac causes.
3. Already surgically closed or otherwise excluded LAA.
4. The LAA anatomy does not accommodate a Closure Device.
5. Known or suspected atrial myxoma.
6. Presence of intracardiac thrombus*.
7. Subjects with a current interatrial baffle or patch, history of atrial septal repair or has an atrial septal defect (ASD) / patent foramen ovale (PFO) device.
8. Subjects with a presence of a mechanical valve prosthesis in any position.
9. Subjects with a myocardial infarction within 90 days prior to enrollment.
10. Subjects had a prior stroke (of any cause, whether ischemic or hemorrhagic) or transient ischemic attack (TIA) within 90 days prior to enrollment.
11. Any planned electrical cardioversion within 30 days following LAAC device implant.
12. Subjects with a known inability to obtain vascular access.
13. Subjects with any contraindication to percutaneous catheterization procedure (e.g., patient size does not accommodate required catheters, ventriculotomy or atriotomy) or congenital abnormalities (severe rotational anomalies of the heart or great vessels) are present.
14. Subjects with any active conditions (e.g. infection, bleeding disorder, unstable angina).
15. Subjects with any contraindications to short term use of anticoagulation therapy for conditions different from atrial fibrillation.
16. Subjects who are pregnant or planning to be pregnant.
17. Subjects with a life expectancy of ≤ 1 year per investigator's opinion.
18. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance must be reviewed by the sponsor to determine eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint (PSE): Device or Procedure Related Serious Adverse Events | 30 days following the index procedure.
  The PSE is the proportion of subjects who experience one or more device- or procedure-related composite serious adverse events (CSAEs) assessed at 30 days following the index procedure.
Primary Efficacy Endpoint (PEE): Acute Treatment Success | Through 30 days
  The PEE is the proportion of subjects with Acute Treatment Success assessed among those receiving ≥ 1 PFA application and who have WATCHMAN device deployment attempted or successfully implanted.

IPD SHARING:
Plan to Share IPD: No